CLINICAL TRIAL: NCT04612959
Title: Effect of Psychosexual Caring Program on Sexual Well-being of Infertile Women: A Randomized Controlled Trial
Brief Title: Effect of Psychosexual Caring Program on Sexual Well-being of Infertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ayse Deliktas Demirci, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AkdenizUniv
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Sexuality; Nursing Caries; Infertility, Female
Keywords: psychoeducation program; infertile women; sexual health; sexual well-being; nursing care
MeSH Terms: conditions — Sexuality; Infertility, Female

STUDY DESIGN:
Intervention Model Description: Randomized controlled double-blind trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The women which participated in the study will not know which group she was in. The data from the groups will be collected by an online survey and the participants will fill form themselves. And data will retreated from the online database by the person who will nt know groups of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosexual care (Experimental): The psychosexual caring program will be conducted online psychoeducation as a group intervention. The program includes four sessions with home assignments and home readings papers.
  Interventions: Other: Psychosexual care
- Standard care (No Intervention): Standard care includes the information given by the nurse about the treatment methods to be applied once.

INTERVENTIONS:
Other: Psychosexual care — The psychosexual caring program includes interventions to promote body awareness, the meaning of sexuality, and marital relationships by gaining communication skills, sexual communication, body knowledge, information about sexual health, and its dimensions.The psychosexual caring program includes psycho-education and sexual counseling.
  Arms: Psychosexual care

SUMMARY:
The present study aims to examine the effect of the psychosexual caring program on the sexual well-being of infertile women.

DETAILED DESCRIPTION:
The study will be conducted with 70 infertile women. The intervention group (n = 35) will consist of infertile women who receive a psychosexual caring program, and the control group will consist of infertile women who receive standard care. Standard care includes the information given by the nurse about the treatment methods to be applied once. A total of 4 interviews will be held in the intervention group. In the first interviews, pre-test data will be taken. The psychosexual caring program will be conducted online as a group intervention. The psychosexual caring program includes interventions to promote body awareness, the meaning of sexuality, and marital relationships by gaining communication skills, sexual communication, body knowledge, information about sexual health, and its dimensions. After online interviews with groups, data will be collected for primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with primary infertility as a result of gynecological evaluation made by experts,
* Planning an assisted reproductive treatment method for women,
* Being active in terms of sexual intercourse,
* Being able to read and write in Turkish,
* Volunteering to participate in the study

Exclusion Criteria:

* Having any known illness related to sexual dysfunction (diabetes, hypertension, heart disease, kidney failure and autoimmune and rheumatic diseases),
* Having a psychiatric diagnosis, •Not having computer or mobile phone and internet access

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
change of sexual function | Data will be collected two times as pre-intervention and immediately post-intervention. After that, change from baseline sexual function at 4 weeks will be assessed.
  Sexual function level of infertile women will be measured by The Female Sexual Function Index (FSFI). Outcome will be assessed based on change of sexual function from baseline at 4 weeks.
change of sexual satisfaction | Data will be collected two times as pre-intervention and immediately post-intervention. After that, change from baseline sexual satisfaction at 4 weeks will be assessed. .
  Sexual satisfaction of infertile women will be determined by using The Sexual Satisfaction Scale for Women. Outcome will be assessed based on change of sexual satisfaction from baseline at 4 weeks.
change of sexual esteem | Data will be collected two times as pre-intervention and immediately post-intervention. After that, change from baseline sexual satisfaction at 4 weeks will be assessed.
  Sexual esteem of infertile women will be measured by The Multidimensional Sexuality Questionnaire-Sexual esteem subscale. Outcome will be assessed based on change of sexual esteem from baseline at 4 weeks.
change of sexual self-efficacy | Data will be collected two times as pre-intervention and immediately post-intervention. After that, change from baseline sexual satisfaction at 4 weeks will be assesed.
  Sexual self-efficacy of infertile women will be measured by Sexual Self-Efficacy Scale.Outcome will be assessed based on change of sexual self-efficacy from baseline at 4 weeks.

SECONDARY OUTCOMES:
change of sense of coherence | Data will be collected two times as pre-intervention and immediately post-intervention. After that, change from baseline sense of coherence at 4 weeks will be assessed.
  Sense of coherence of infertile women will be determined by Sense of Coherence Scale.Outcome will be assessed based on change of sense of coherence from baseline at 4 weeks.
change of depression | Data will be collected two times as pre-intervention and immediately post-intervention. After that, change from baseline depression at 4 weeks will be assessed .
  Depression level of infertile women will be measured by Beck Depression scale.Outcome will be assessed based on change of depression from baseline at 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kamile Kabukcuoglu, Study Director — Akdeniz University; Ayse Deliktas Demirci, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aydin S, Beji NK. Sexual function in infertile couples and the role of infertility counselor. Journal of Education and Research in Nursing. 2013; 10(2): 8-14.
- [Background] Mendonca CR, Arruda JT, Noll M, Campoli PMO, Amaral WND. Sexual dysfunction in infertile women: A systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2017 Aug;215:153-163. doi: 10.1016/j.ejogrb.2017.06.013. Epub 2017 Jun 7. PMID 28628848
- [Background] Evans DT. Promoting sexual health and wellbeing: the role of the nurse. Nurs Stand. 2013 Nov 6-12;28(10):53-7; quiz 60. doi: 10.7748/ns2013.11.28.10.53.e7654. PMID 24191835
- [Background] Martin, K. M., Woodgate, R. L. 2017. "Concept analysis: The holistic nature of sexual well-being", Sexual and Relationship Therapy, 1-15.
- [Background] Read SC, Carrier ME, Boucher ME, Whitley R, Bond S, Zelkowitz P. Psychosocial services for couples in infertility treatment: what do couples really want? Patient Educ Couns. 2014 Mar;94(3):390-5. doi: 10.1016/j.pec.2013.10.025. Epub 2013 Nov 5. PMID 24290241